CLINICAL TRIAL: NCT06937606
Title: A Randomized, Controlled Trial to Increase Self-compassion and Decrease Caregiving Fatigue in Group Leaders of a Support Group for Women After Cancer (GLOW) - an Adaption of the Mindful Self-Compassion Program for Healthcare Communities
Brief Title: Decrease Caregiving Fatigue in Group Leaders of a Support Group for Women After Cancer
Acronym: GLOW
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Robert Bosch Medical Center (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Claudia Loeffler, PD Dr. med., Senior physician, Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 171/23-am
Record Dates: First submitted 2024-09-23; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Caregiver Burden
Keywords: self-compassion training; cancer care; empathy fatigue; burnout; resilience
MeSH Terms: conditions — Caregiver Burden; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-compassion training (Experimental): Online group intervention: led by a certified mindfulness teacher for mindful self-compassion and additional qualification in self-compassion in healthcare communities (duration: 6 weekly appointments of 90 min each);
  Interventions: Behavioral: Self-compassion training
- waiting list control (No Intervention): waiting list control

INTERVENTIONS:
Behavioral: Self-compassion training — Online group intervention: led by a certified mindfulness teacher for mindful self-compassion and additional qualification in self-compassion in healthcare communities (duration: 6 weekly appointments of 90 min each);
  Arms: Self-compassion training

SUMMARY:
This exploratory study aims to evaluate the effect of a self-compassion training developed for health professionals on leaders of self-help groups.

Hypothesis/primary goal: An online group intervention adapted from the "Self-compassion for health-care communities program" validated for health professionals leads to an increase in self-compassion among leaders of cancer self-help groups. Secondary goals: level of self-compassion at the end of the course as a mediator for therapeutic variables after 6 weeks, decrease in caregiver fatigue, secondary traumatic stress/burnout risk, personal distress and sick leave, decrease in fears of self-compassion/compassion for others; increase in mindfulness, self-efficacy, compassion for others and resilience; direct costs; safety;

Intervention:

Online group intervention: led by a certified mindfulness teacher for Mindful Self-Compassion and additional qualification in Self-Compassion in Healthcare Communities (duration: 6 weekly appointments of 90 min each); control intervention: waiting group

ELIGIBILITY:
Inclusion Criteria:

* Group leaders of a self-help group for cancer patients
* written informed consent

Exclusion Criteria:

* Medical or mental condition that, in the opinion of the investigator, does not allow the participant to take part in the study or to provide a legally valid signature of the informed consent (e.g. insufficiently controlled pre-existing mental illness or post-traumatic stress disorder)
* Lack of willingness to store and share personal health data as part of the protocol
* Participation in another mindfulness study
* Lack of knowledge of German

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
self-compassion as assessed by Self-compassion scale in german version (SCS-D) | 6 weeks after baseline
  Determining self-compassion after the intervention by means of a confirmatory test for group differences in the primary endpoint according to the ITT principle using a linear regression model; instrument: SCS-D

SECONDARY OUTCOMES:
Decrease in compassion fatigue as assessed by ProQoL | 12 weeks after baseline
  Professional Quality of Life (ProQOL) is intended for any helper - health care professionals, social service workers, teachers, attorneys, emergency response, etc. Understanding the positive and negative aspects of helping those who experience trauma and suffering can improve your ability to help them and your ability to keep your own balance.
secondary traumatic stress/burnout risk as assesd by ProQoL | 12 weeks after baseline
  Professional Quality of Life (ProQOL) is intended for any helper - health care professionals, social service workers, teachers, attorneys, emergency response, etc. Understanding the positive and negative aspects of helping those who experience trauma and suffering can improve your ability to help them and your ability to keep your own balance.
personal distress (PSS-10) | 12 weeks after baseline
  The Perceived Stress Scale (PSS-10) is a 10-item questionnaire originally developed by Cohen et al. (1983) widely used to assess stress levels in young people and adults aged 12 and above. It evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the previous month.
decrease in fears of self-compassion (FCS) | 12 weeks after baseline
  The FCS-A assesses fear of compassion for self, fear of compassion for others, and fear of compassion from others and. It identifies barriers to giving compassion to oneself (15 items), to others (10 items), and receiving compassion from others (13 items). The items are rated on a five-point Likert scale (0 = Don't agree at all, 4 = Completely agree). The higher the score, the greater the one's fears, blocks and resistances to compassion.
compassion for others (COS-7) | 12 weeks after baseline
  The questionnaire uses a 7 point Likert scale ranging from 1 (not at all true of me) to 7 (very true of me) to capture levels of compassion. Total scores are derived by averaging all item scores. Higher total scores indicate higher levels of compassion for others (strangers). https://doi.org/10.1007/s12144-020-01344-5
increase in mindfulness (FFMQ) | 12 weeks after baseline
  The Five Facet Mindfulness Questionnaire (FFMQ-15) is a 15 question self-report scale that measures mindfulness with regards to thoughts, experiences, and actions in daily life (Baer, Carmody, & Hunsinger, 2012).
increase in self-efficacy (SWE) | 12 weeks after baseline
  The scales can be used to measure beliefs about subjective controllability and competence expectations in various demanding situations, namely at school, in higher education, and in everyday life. The method is primarily intended for use in scientific research.
  Jerusalem, M. & Schwarzer, R. (1981). "Selbstwirksamkeit". WIRK. In R. Schwarzer (Hrsg.) (1986), Skalen zur Befindlichkeit und Persönlichkeit (Forschungsbericht 5. S. 15-28). Berlin: Freie Universität, Institut für Psychologie.
increase in resilience (BRS) | 12 weeks after baseline
  The BRS is a reliable means of assessing resilience as the ability to bounce back or recover from stress and may provide unique and important information. The BRS consists of six items. Items 1, 3, and 5 are phrased positively, while items 2, 4, and 6 are phrased negatively. The BRS is evaluated by recoding items 2, 4, and 6 and calculating the mean value of the six items.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Löffler, PD Dr. med., Principal Investigator — Medizinische klinik und Poliklinik II
Locations (1):
- Comprehensive Cancer Center Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No